CLINICAL TRIAL: NCT06134206
Title: Evaluation of the Feasibility of Measuring Chronic Subdural Hematoma Thickness Via Trans-burrhole Ultrasound
Brief Title: Burr Hole Ultrasound Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC Nr. 1054/2022
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Subdural Hematoma
Keywords: Burr hole; Ultrasound; Trans-burr hole; TBUS; Sonography; Chronic Subdural hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Intervention Model Description: 1 Group of 20 patients who all underwent the same examination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Burr hole sonography (Experimental): Patients within this arm (only arm of the study) undergo burr hole sonography
  Interventions: Diagnostic Test: Trans-burr hole ultrasound

INTERVENTIONS:
Diagnostic Test: Trans-burr hole ultrasound — All ultrasound examinations were conducted alongside the routine postoperative CT scan between 3-7 days postoperatively. To minimize potential influences of the patient's head position on the distribution and thickness of the subdural fluid, we first carried out the CT scan with the patient and their head in a supine position. Immediately after the CT scan, the patient remained on the same examination bed, and burr hole ultrasound was performed in the identical supine position. The burr hole was centered in the image, with the outer table surrounding the burr hole displayed as a horizontal line. The content of the burr hole could be differentiated by its higher echogenicity from the subdural residual hematoma or residual fluid. The brain's surface and overlying leptomeninges, however, displayed higher echogenicity compared to the subdural fluid. The subdural hematoma's thickness was measured at its maximum extent.
  Other Names: TBUS; Trans-burr hole sonography; burr hole sonography; burr hole ultrasound

SUMMARY:
Chronic subdural hematoma (CSDH) is commonly managed through burr hole evacuation. This study evaluates the feasibility of trans burr hole sonography as an alternative postoperative imaging modality.

A pilot study on 20 patients who underwent burr hole surgery for CSDH was therefore planned. Postoperative imaging included both CT and sonographic examinations through the burr hole. We assessed the ability to measure residual subdural fluid thickness sonographically compared to CT.

ELIGIBILITY:
Inclusion Criteria:

* Burr hole surgery due to chronic subdural hematoma
* Routine performance of an computed tomography scan within 3-7 days postoperative
* Ability to give informed consent

Exclusion Criteria:

* Performance of prior craniotomy
* Performance of prior revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
cSDH thickness | 1 measurement on day 3-7 postoperative
  maximum extent of the hematoma (chronic subdural hematoma, CSDH) thickness under the burr hole in axial and coronal plane

CONTACTS AND LOCATIONS:
Overall Officials: Harald Stefanits, MD, PhD, Principal Investigator — Department of Neurosurgery, Kepler University Hospital Linz, Austria
Locations (1):
- Department of Neurosurgery, Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aspalter S, Gmeiner M, Gasser S, Sonnberger M, Stroh N, Rauch P, Gruber A, Stefanits H. Feasibility, Clinical Potential, and Limitations of Trans-Burr Hole Ultrasound for Postoperative Evaluation of Chronic Subdural Hematoma: A Prospective Pilot Study. Neurosurgery. 2024 Oct 1;95(4):924-931. doi: 10.1227/neu.0000000000002957. Epub 2024 Apr 22. PMID 38647289